CLINICAL TRIAL: NCT04563585
Title: Position Differences and Physical Performance Among Female Team Handball Players
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Cyprus International University (Other)
Responsible Party: Principal Investigator, caglar soylu, Çağlar Soylu, Ankara Yildirim Beyazıt University
Other Study IDs: 2020-242
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Handball Players; Position Differences; Physical Performance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Muscle strength: Maximal voluntary isometric (MVIC) knee flexion and extension strength were measured using a handheld dynamometer (HDD) (Lafayette Instrument Company, Lafayette, IN).
- Lower Extremity Vertical Power: Lower extremity vertical power was identified through the use of the VertiMetric (Lafayette Instrument Company, Lafayette, IN) according to protocols suggested by Ambegaonkar et al.
- Trunk Extension Endurance: Trunk extension endurance was measured using the Biering-Sorensen test as previously described
- Upper Limb Performance: The Davies test (DT) was used to assess upper body agility and stabilization.The Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) was utilized to assess shoulder performance function and stability according to protocol suggested by Goldbeck and Davies.
- Lower Limb Performance: The Shark Skill Test (SST) was developed in order to assess lower extremity agility and neuromuscular control.

SUMMARY:
Our study was conducted to compare the physical performances of the upper extremity and lower extremity of handball players according to the positions they played.

In this cross-sectional study, a total of 39 elite female handball players with at least of 5 years playing experience were tested.Maximal voluntary isometric (MVIC) knee flexion and extension strength were measured using a handheld dynamometer (HDD) (Lafayette Instrument Company, Lafayette, IN). Lower extremity vertical power was identified through the use of the VertiMetric (Lafayette Instrument Company, Lafayette, IN) according to protocols suggested by Ambegaonkar et al. Trunk extension endurance was measured using the Biering-Sorensen test as previously described.The Davies test (DT) was used to assess upper body agility and stabilization.The Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) was utilized to assess shoulder performance function and stability according to protocol suggested by Goldbeck and Davies.The Shark Skill Test (SST) was developed in order to assess lower extremity agility and neuromuscular control.

ELIGIBILITY:
All athletes were asymptomatic and had passed medical examinations prior to inclusion and participation in the study. Exclusion criteria included history of injury or surgery that may affect their lower and upper limbs and any lower and upper limb injuries within the last three months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In this cross-sectional study, a total of 39 elite female handball players with at least of 5 years playing experience were tested. Player positions were identified for each athlete by their coaches or by self-report as: goalkeepers, centres, pivots, or wing players. All of them were playing in the premier Turkish professional handball league.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | 2 weeks
  Maximal voluntary isometric (MVIC) knee flexion and extension strength were measured using a handheld dynamometer (HDD) (Lafayette Instrument Company, Lafayette, IN).
Lower Extremity Vertical Power | 2 weeks
  Lower extremity vertical power was identified through the use of the VertiMetric (Lafayette Instrument Company, Lafayette, IN) according to protocols suggested by Ambegaonkar et al.
Trunk Extension Endurance | 2 weeks
  Trunk extension endurance was measured using the Biering-Sorensen test as previously described.
Upper Limb Performance | 2 weeks
  The Davies test (DT) was used to assess upper body agility and stabilization.The Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) was utilized to assess shoulder performance function and stability according to protocol suggested by Goldbeck and Davies.
Lower Limb Performance | 2 weeks
  The Shark Skill Test (SST) was developed in order to assess lower extremity agility and neuromuscular control.

CONTACTS AND LOCATIONS:
Overall Officials: Bünyamin Haksever, PhD, Principal Investigator — Cyprus International University
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No